CLINICAL TRIAL: NCT05655858
Title: Observational Study of Allergic Rhinitis in Children
Acronym: ORACLE
Status: Completed | Type: Observational
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-A01596-37
Record Dates: First submitted 2022-12-01; First posted 2022-12-19 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Management of allergic rhinitis — Collection of patient data in real-life

SUMMARY:
Observational, cross-sectional, prospective, multicentric study in France with private paediatricians to describe the management of allergic rhinitis in children.

DETAILED DESCRIPTION:
Data collected about diagnostic, comorbidities, clinical history, management of allergic rhinitis using a patient paper case report form. There is only one visit per patient and investigators can include up to 20 patients.

ELIGIBILITY:
Inclusion Criteria:

* Under 18 years of age
* With allergic rhinitis
* Who's representative of the parental authority did not object to his child's participation after oral and written information and who agrees to participate

Exclusion Criteria:

* Child or adolescent opposed to participate or collect his personal data

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 1000 patients aged 2 to 18 years old with allergic rhinitis
Sampling Method: Probability Sample
Enrollment: 1004 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2024-03-03 (Actual); Study Completion 2024-03-03 (Actual)

PRIMARY OUTCOMES:
Proportion of children over 2 years of age with allergic rhinitis eligible for allergic immunotherapy | 1 year
  Descriptive analysis : evaluation with data collected in the case report form about allergic rhinitis

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Necker-Enfants malades - AP-HP Service de Pneumologie et Allergologie Pédiatriques, Paris, France

IPD SHARING:
Plan to Share IPD: No